CLINICAL TRIAL: NCT06103448
Title: Prediction of the Risks of Cardiovascular Mortality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jan Evangelista Purkyne University (Other)
Responsible Party: Principal Investigator, Iva Volešová, Clinical Instructor, Jan Evangelista Purkyne University
Other Study IDs: IGA-FZS-2023-6
Record Dates: First submitted 2023-10-11; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases; Cardiovascular Morbidity; Stroke; Embolism; Cardiac Arrest
Keywords: ankle-brachial index; cardiovascular mortality; prevention
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Embolism; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ankle-brachial index - system 100 — Measurement of ankle brachial index on all four limbs, drawing three blood drops for point of care (POC) cholesterol meter and one drop of blood for POC glucometer
  Other Names: Point of care cholesterol meter by Lux and point of care Glucometers

SUMMARY:
Monitoring risks of cardiovascular diseases in working population (18 - 65 years old) by monitoring their BMI, ankle-brachial index with pulse wave velocity, cholesterol and glycemia.

DETAILED DESCRIPTION:
Monitoring working population in their workplace by measuring their ankle-brachial index with pulse wave velocity, BMI, glycemia and cholesterol. Putting acquired data in correlation to their work habits, type of employment, work demands, job type, activity levels. Trying to find common predictors of cardiovascular disease. All assessed subjects must understand written and spoken Czech, must be employed in a company that consents with our data collections, must be older than 18 year old, doesn't have any bleeding disorder, doesn't have deep vein thrombosis (as it produces inaccurate data with ankle brachial index). Study will be conducted in Ustecky Region in the Czech Republic on approximately 200 subjects.

ELIGIBILITY:
Inclusion Criteria:

* employed in Ustecky Region Czech Republic
* adult
* understands spoken and written Czech
* consents with assessment
* works in a company that consents to assessments of their employees

Exclusion Criteria:

* deep vein thrombosis
* not currently employed
* on sick leave
* bleeding disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Working individuals with employment contract in Ustecky Region, that are able to consent to assessment, are adults and understand written and spoken Czech language. Random companies from Ustecky region will be approached with the opportunity to participate.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Detection of glycemia, HDL, LDL and triacylglyceride levels | 5 minutes
  Glycemia, HDL, LDL and triacylglyceride levels (mmol/l) will be measured from drops of blood by point-of-care analysers
Body composition | 3 minutes
  Using body composition scale the following markers will be counted: bone mass, body fat, muscle mass, water levels. All results will be in %
Ankle-brachial index | 2 minutes
  Ankle-brachial index (no unit) using ABI-system-100 will be counted from blood pressure measured in all four limbs (mmHg)
Ankle brachial pulse wave velocity (baPWV) and carotid femoral pulse wave velocity (cfPWV) | 2 minutes
  baPWV and cfPWV will be measure by ABI-system-100 (m/s)
Weight | 1 minute
  measured by body composition scale (kg)
Height | 1 minute
  measured by tailor tape measure (m)

SECONDARY OUTCOMES:
BMI | 2 minutes
  BMI (kg/m^2) will be counted from weight (kg) and height (m)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jan Evangelista Purkyně, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: No